CLINICAL TRIAL: NCT04461171
Title: Enhanced Recovery After Surgery in Extremity Sarcoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joshua Lawrenz (Other)
Responsible Party: Sponsor-Investigator, Joshua Lawrenz, Principal Investigator, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VICC SAR 2020
Record Dates: First submitted 2020-06-10; First posted 2020-07-08 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Sarcoma
Keywords: Enhanced Recovery After Surgery
MeSH Terms: conditions — Sarcoma | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Intervention Model Description: Two-group, prospective, consecutively enrolled, comparative non-randomized trial (N = 120) is to determine the feasibility and efficacy of implementing an enhanced recovery after surgery (ERAS) pain management pathway to patients undergoing surgical treatment for an extremity sarcoma.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS (Experimental): Administration of a perioperative non-narcotic, multimodal pain management pathway.
  Interventions: Procedure: Enhanced Recovery After Surgery
- Non-ERAS (Conventional) (No Intervention): Administration of a conventional perioperative pain management pathway that consists of both narcotic and non-narcotic pain medications.

INTERVENTIONS:
Procedure: Enhanced Recovery After Surgery — Undergo an enhanced recovery after surgery program
  Arms: ERAS

SUMMARY:
The purpose of this study is to demonstrate the efficacy of implementing the enhanced recovery after surgery (ERAS) pathway in a prospective manner to patients undergoing surgical treatment for extremity sarcoma.

DETAILED DESCRIPTION:
Specifically, the focus of this study will be regarding the administration of a perioperative non-narcotic, multimodal pain management pathway. Primary endpoints collected with be short-term patient reported outcomes (pain scores [PROMIS] and [QoR-15]), limb function scores [MSTS], and key clinical outcomes (hospital length of stay, opioid requirements/prescribing data and perioperative complications).

ELIGIBILITY:
Inclusion Criteria:

* Any patient at Vanderbilt University Medical Center treated with surgical excision of a suspected extremity sarcoma
* Adult patients >17 years of age
* Patients of all preoperative opioid status (naïve or dependent)

Exclusion Criteria:

* Patients treated non-operatively
* Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pain scores | 3 months
  Measured by Quality of Recovery questionnaire (QoR-15) scale = 0-10 (0=none of the time and 10 = all of the time)
Pain scores | 3 months
  Measured by Patient-Reported Outcomes Measurement Information System (PROMIS-29 Profile v2.0) Score 1-5 (1 being worst and 5 being best)
Limb function | 3 months
  Measured by Musculoskeletal Tumor Society scoring system (MSTS) scored from 0-5 (5 being best and 0 being worst)
Clinical outcomes - length of hospital stay | 3 months
  Measured by the number of days in the hospital
Clinical outcomes - opioid requirements | 3 months
  Measured by the amount of opioids consumed
Clinical outcomes - perioperative complications (e.g. wound complications and 30-day readmission) | 3 months
  Measured by the number of perioperative complications reported

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Lawrenz, MD, Principal Investigator — Vanderbilt Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT04461171/ICF_000.pdf